CLINICAL TRIAL: NCT04866745
Title: Effectiveness of Magnetotherapy and Microwaves Combined With Therapeutic Exercise in Patients With Knee Osteoarthritis.
Brief Title: Magnetotherapy Versus Microwave Combined With Exercise for Knee Osteoarthritis.
Acronym: MT-MW-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Centro de Salud Talavera Centro y Centro de Salud La Algodonera. (Unknown); Clínica Radiodiagnóstico Marazuela (Unknown); Empresa Helios Electromedicina S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: magneto-gifto
Record Dates: First submitted 2021-03-25; First posted 2021-04-30 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis; Pain
Keywords: Knee osteoarthritis; Pain; Function; Phychosocial
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Magnetic Field Therapy; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Double-blinded, sham-controlled, randomized clinical trial.
Who Masked: Participant, Investigator
Masking Description: The assignment to the MT and MT placebo group will be only known by the technician from the external device manufacturer who programs the coded MT equipment. The coded MT equipment will be programmed in such a way that the physical therapist that applies the intervention will enter the code for each participant without knowing the group to which the patient is assigned. Therefore, the therapists that apply the intervention will only know the assignment to the MW group. For the blinding of the subjects, the same protocol will be followed in the placebo treatment as in the experimental group (number of sessions, application area, and device). The researchers who perform the recruitment, the participants, the researcher who will perform the assessments and the analysis of the data, and the therapists who will apply the exercise program will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Magnetotherapy plus exercise (Experimental): The patients will receive a total of 12 sessions, 3 sessions per week of magnetotherapy. The duration of treatment will be 20 minutes with a magnetic field frequency of 50Hz and a power of 100 Gauss.
  After the magnetotherapy treatment, the patient will have to perform 12 sessions, 3 sessions per week of a program of therapeutic exercise with a duration of 25 minutes. This exercise program will be the same in the microwave and sham groups.
  Interventions: Device: Magnetotherapy plus exercise
- Sham Magnetotherapy plus exercise (Placebo Comparator): The patients will receive a total of 12 sessions, 3 sessions per week of sham magnetotherapy. For the simulated/sham magnetotherapy group, it will be applied in the same way as the real MT group, but the equipment will be programmed to apply 0 Gauss. The physiotherapist performing the application will not have access to the magnetotherapy parameters on the display of the device, but will only have to enter the code. After the application of sham magnetotherapy, the patient will have to perform a program of therapeutic exercise.
  Interventions: Device: Sham Magnetotherapy plus exercise
- Microwave plus exercise (Active Comparator): The patients will receive a total of 12 sessions, 3 sessions per week of microwave therapy. The duration of the session will be 20 minutes, 10 minutes on the anterior side and 10 minutes on the posterior side of the joint in case of unilateral knee osteoarthritis. In the case of bilateral knee osteoarthritis, the MW will be applied 20 minutes over the anterosuperior side of both knees. After the microwave session, the patient will have to perform a program of therapeutic exercise.
  Interventions: Device: Microwave plus exercise

INTERVENTIONS:
Device: Magnetotherapy plus exercise — The VARIMAG-4E magnetotherapy device will be used. It is a pulsed radiofrequency energy device. The device has a voltage of 220V, 4 amps of intensity, 50 Hz of frequency and a maximum power of 100 Gauss. For the active treatment application, the patient will be in supine position and will introduce both knees in the 50 cm coil in case of bilateral knee osteoarthritis. In the case of unilateral knee osteoarthritis, the affected knee will be introduced in the 30cm coil. The duration of the treatment will be 20 minutes, the frequency administered will be 50 Hz and a power of 100 Gauss.
  Other Names: Magnetotherapy, VARIMAG-4E.
  Arms: Magnetotherapy plus exercise
Device: Microwave plus exercise — The application of deep heating therapy will be with the patient in a sitting position. The VARITRON 250-EP microwave device will be used with a frequency of 2450 MHz and a maximum output power of 250W. In the case of unilateral knee osteoarthritis, the circular applicator with a diameter of 170mm will be placed approximately 15 cm from the knee. The duration of the session will be 20 minutes, 10 minutes over the internal face and 10 minutes over the external face of the knee. In the case of bilateral knee osteoarthritis, the large lumbar applicator will be placed approximately 15 cm from the anterosuperior face of both knees for 20 minutes. The patient will have to perceive a moderate heat sensation.
  Other Names: Deep heating therapy, VARITRON 250-EP.
  Arms: Microwave plus exercise
Device: Sham Magnetotherapy plus exercise — The protocol and device will be the same in the active/placebo treatment. The sham device does not emit an electromagnetic field. The energy from the active device is not felt by the user, and the active device cannot be distinguished in any way from the placebo device.
  Other Names: Sham Magnetotherapy, VARIMAG-4E.
  Arms: Sham Magnetotherapy plus exercise

SUMMARY:
The high prevalence of knee osteoarthritis and the absence of well-defined protocols for the application of Magnetotherapy (MT), makes it necessary to investigate the effect of this therapy on patients with knee osteoarthritis. Furthermore, no studies are comparing the effectiveness of the two interventions proposed in this project (MT) and microwaves (MW), which are routinely applied in clinical practice, without solid scientific evidence to justify their use.

The purpose of the present clinical trial is to compare MT with MW both combined with a therapeutic exercise program in patients with painful knee osteoarthritis and its influence on pain and function.

DETAILED DESCRIPTION:
This study is a double-blinded, sham-controlled, randomized clinical trial whose main objective is to investigate the effect on pain and function in people with moderate knee osteoarthritis of the intervention with Magnetotherapy (MT) combined with an exercise program compared to microwave (MW) application combined with an exercise program and to MT placebo combined with an exercise program. The study will take place at several centers of primary healthcare centers in Spain. After receiving the approval of the Ethics and Clinical Research Committee of Talavera de la Reina Hospital (Toledo). It is proposed to perform the study between May 2021 to May 2022.

The secondary objectives are:

* To investigate the effect of intervention with MT and MW plus exercise on quality of life and psychosocial factors of pain in people with osteoarthritis of the knee.
* To evaluate the effect of both interventions on knee joint kinematics and range of motion and lower limb strength.
* To evaluate the success of the blinding method of participants and professionals.
* To measure the possible adverse effects of the application of MT and MW in patients with moderate osteoarthritis of the knee.

The participants will be randomly assigned in three groups:

* Group A: Magnetotherapy combined plus exercise program.
* Group B: Sham magnetotherapy plus exercise program.
* Group C: Microwaves combined plus exercise program.

A minimum of 60 adults, older than 45 years old, diagnosed with osteoarthritis of the knee who meet the inclusion criteria will be recruited by voluntary admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 45 years old
* Unilateral or bilateral knee osteoarthritis.
* Kellgren and Lawrence (K-L) grade II or III.
* Visual analog scale (VAS) greater than 40mm.
* Affectation of more than one year of evolution.
* Sign and understand the informed consent form.

Exclusion Criteria:

* Secondary cause osteoarthritis
* History of uncontrolled metabolic diseases.
* Decompensated or uncontrolled pathologies
* Tumor processes.
* Collagenopathies and neurological diseases.
* Changes in medication or invasive treatments at least 1 month prior to treatment.
* Receiving physiotherapy treatment or having received it one month prior to the start of the osteoarthritis study.
* Patients with alterations in thermal sensitivity.
* Pacemaker
* Skin alterations (recent wounds or burns).
* Knee prosthesis
* Thrombophlebitis

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Change in knee pain | Change from baseline at 4 weeks, 1 month and 4 months after intervention.
  The knee pain perceived in motion and at rest will be measured with the standard 10 cm Visual Analog Scale (VAS). It will be expressed in mm. Being the value 0 "no pain" and the value 10 "worst pain".
Change in function | Change from baseline at 4 weeks, 1 month and 4 months after intervention.
  Physical function, pain, and stiffness will be measured with the Western Ontario and McMaster Universities Arthritis Index (WOMAC-24). It is a self-administered questionnaire consisting of 24 items divided into 3 subscales. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Daily knee pain | Before each treatment session. 3 sessions per week (total 4 weeks)
  The daily level of knee pain will be measured before every session of treatment using a standard 10 cm Visual Analog Scale (VAS). It will be expressed in mm. The value 0 will be the best and 10 the worst functionality.
Daily level of functionality | Before each treatment session (during 4 weeks)
  The level of functionality will be measured before every session of treatment using a standard 10 cm Visual Analog Scale (VAS). It will be expressed in mm. The value 0 will be the best and 10 the worst functionality.
Daily quality of sleep | Before each treatment session (during 4 weeks)
  The quality of sleep will be measured before every session of treatment using a standard 10 cm Visual Analog Scale (VAS). It will be expressed in mm. The value 0 will be the best and 10 the worst.
Daily intake of oral non-opioid analgesic medication | Before each treatment session (during 4 weeks)
  Daily intake of oral non-opioid analgesic medication (number of pills per day) during the 24 hours interval before each treatment session being the value 0 the best and 10 the worst.
Change in balance and fall risk | Mean differences from baseline at 4 weeks, 1 month and 4 months after intervention.
  Test timed up and go (TUG) will be expressed in seconds. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down. The test will be performed 3 times. The mean of the three tests will be used. Less time performing this test indicates better mobility.

SECONDARY OUTCOMES:
Change in patient quality of life | Index change from baseline at 4 weeks, 1 month and 4 months after intervention.
  The European Quality of life 5 Dimensions (EuroQoL 5D-5L) is a questionnaire that evaluates the generic quality of life measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each health state is usually represented using a 5-digit number (profile) where 11111 indicates perfect health and 55555 the worst health state.
Change in lower limb strength | Mean difference from baseline at 4 weeks, 1 month and 4 months after intervention.
  Maximal isometrical knee extension and flexion strength will be measure with a hand dynamometer and will be expressed in Kgs. The researcher will perform three measurements and the final result will be the average of the three.
Blinding assesment | Post treatment at 4 weeks
  The success of participant and assessor blinding will be evaluated through a questionnaire after each intervention with five questions: (1) "Strongly believe the applied intervention is new treatment"; (2) "Somewhat believe the applied intervention is new treatment"; (3) "Somewhat believe the applied intervention is a placebo", (4) "Strongly believe the applied intervention is a placebo", or (5) "Do not know".
Number of participants with adverse effects | Post each treatment session (during 4 weeks)
  The number of participants who suffered adverse effects will be reported by the researcher (for example skin erythema, rush, or itching...).
Change in knee range of motion | Mean difference from baseline at 4 weeks, 1 month and 4 months after intervention.
  Knee active and passive range of motion will be measure with the WERIUM sensors. It will be expressed in degrees. The mean of 3 movements of flexion and extension will be calculated.
Change in perceived generic health status | Change from baseline at 4 weeks, 1 month and 4 months after intervention.
  The European Quality of life 5 Dimensions (EuroQoL 5D-5L) questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Doses of analgesic and antidepressant medication | Change from baseline at 4 weeks.
  The doses of analgesic and antidepressant medication will be recorded at baseline.
  Taking into account the therapeutic steps of the World Health Organization and the dosage, 4 values will be established concerning the basal state: "increases, decreases, it is eliminated or it is maintained".

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Avendaño Coy, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Yes
Congress presentation in a poster format Publication in a scientific journal Social media
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 01/01/2023. The data will be published in a scientific journal